CLINICAL TRIAL: NCT05264870
Title: Norepinephrine as Hemodynamic Maintenance in Caesarian Delivery Under Spinal Anesthesia
Brief Title: Norepinephrine in Caesarian Section
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: patient inclusion is too difficult
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, Hilde Coppejans, Principle Investigator, University Hospital, Antwerp
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 002105
Record Dates: First submitted 2022-02-22; First posted 2022-03-03 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Cesarean Section Complications; Hemodynamic Instability; Foetal Stress
MeSH Terms: interventions — Norepinephrine

STUDY DESIGN:
Intervention Model Description: Norepinephrine infusion is given for treatment of postspinal hypotension in treatment group A and B
Who Masked: Participant, Outcomes Assessor
Masking Description: Both the patient and the observant/study physician are fully blinded. Randomization, preparation of study medication and administration of CSE anesthesia is performed by a protocol trained anesthesiologist. He or she is further excluded to any other study related intervention. A second protocol trained anesthetist comes in and will adapt the norepinephrine infusion according to the needs of the patient. He will do routine care observations and interventions until end of surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Active Comparator): combined spinal epidural anesthesia (CSE) with 7,5mg hyperbaric Marcaine and 2,5mcg Sufentanil
  Interventions: Drug: Norepinephrine
- Group B (Active Comparator): combined spinal epidural anesthesia (CSE) anesthesia with 10mg hyperbaric Marcaine and 2,5mcg Sufentanil
  Interventions: Drug: Norepinephrine

INTERVENTIONS:
Drug: Norepinephrine — treatment of postspinal hypotension
  Arms: Group A
Drug: Norepinephrine — treatment of postspinal hypotension
  Arms: Group B

SUMMARY:
Postspinal hypotension is a frequent maternal complication in caesarian delivery under neuraxial anesthesia which is most commonly treated with the administration of phenylephrine infusion. In this trial, postspinal hypotension will be treated with norepinephrine. The main objective is to examine the pharmacodynamic and biochemical effect of norepinephrine both on mother and newborn.

DETAILED DESCRIPTION:
Patients scheduled for routine elective cesarean section under combined spinal epidural anesthesia (CSE)will be enrolled in this double-blind, randomized controlled trial, As standard of care for cesarean section procedure, a preoperative anesthetic consultation is performed. If the patient is eligible for enrollment, she will be provided with detailed information regarding the study and asked to sign Informed Consent. Participants are allocated to one of two groups: Group A will receive a CSE anesthesia with 7,5 milligrams (mg)hyperbaric Marcaine and 2,5 microgram (mcg)Sufentanil.

Group B will receive a CSE anesthesia as well with 10 mg hyperbaric Marcaine and 2,5 mcg Sufentanil. At the University Hospital Antwerp, Group A is standard of care for cesarean section. In case of insufficient pain relief an extra bolus of local anesthesia through the epidural catheter can be administered in both groups. In this trial we use a double blinding principle. Both the patient and the observant/study physician are fully blinded. To maintain blinding of the study, two anesthesiologists are involved in this trial. The first anesthesiologist will perform randomization by means of Redcap software and will prepare study medication according to allocation to group A or B just before start of spinal anesthesia. He /she is responsible for the placement of neuraxial block and the spinal epidural catheter. As part of routine care anesthesia an intravenous line with 500 milliliter (ml) Plasmalyte (minimal 20 Gauche catheter) will be established in both groups . Standard monitoring (blood pressure, Electrocardiogram and Oxygen saturation) will be applied.

A baseline systolic blood pressure will be measured as a mean of 3 consecutive measurements before start of CSE and is defined as baseline blood pressure.

Blood pressure will be measured every 1 minute. To maintain normotension during the procedure a continuous infusion of norepinephrine will be given at 15 milliliter/hour through the peripheral intravenous (IV)catheter in both groups. Therefore a solution of norepinephrine in a concentration of 10mcg/ml in a 50ml syringe is prepared and connected to the peripheral IV line, most proximal to the IV catheter. A combined spinal epidural puncture will be performed in the sitting position at the level of Lumbal (L)2-L3 or L3-L4 with a CSE needle set (18 Gauge Tuohy needle, 27 Gauge pencil point needle, 18 gauge catheter, Braun).

After placing the 18-gauge Tuohy needle in the epidural space, confirmed by loss of resistance with natriumchloride (NaCl) 0,9 percent (%), the spinal 27-gauge pencil point needle is advanced until it reaches the subarachnoidal space. Once the wright needle tip position is confirmed by back flow of cerebrospinal fluid (CSF), the local anesthetic solution will be injected in 15 seconds with the spinal needle orifice facing cephalad. Immediate after injection the epidural catheter will be inserted and placed at a distance of 5 cm beyond the Tuohy needle tip. Afterwards the patient is turned to the supine position A left lateral tilt (30%) will be applied to the operating table.

The Trendelenburg position of the table may be changed from -15 degree(°) to 15 ° table if necessary according to the anaesthetist in charge who is blinded for the appointed study group. In the unusual case of insufficient analgesia a single top-up dose of 5ml lidocaine 2% can be given through the epidural catheter. The bladder will be catheterized after spinal puncture. The start time of the recordings (T0) is the injection of the spinal anesthesia. At this moment we start the continuous infusion of norepinephrine. The anesthesiologist who performed the spinal anesthesia will leave the operating room and is replaced by a protocol trained second anesthesiologist to maintain blinding. The observer is always unaware of the appointed study group. He/she will titrate the continuous infusion of norepinephrine. In case of hypotension, defined as a decrease of 10% (more or equal) from baseline systolic arterial pressure, or an absolute value lower than( <) 100 mmHg, norepinephrine infusion will be increased with 2ml/hr each time with a maximum of 30ml/hr. Patients receive no extra volume loading besides a standard crystalloid infusion at a continuous rate of 80ml/u.

In case of hypertension, systolic blood pressure of more than 10% above baseline, the infusion will be lowered by 2ml/hr. Observation of vital parameters will be continued until safe delivery of the baby. Blood samples from the umbilical cord immediately after birth is part of standard of care.

With a non-inferiority margin of 0,05 we will need a sample size of 39 patients per group. Data will be collected using Redcap software to maximize transparency. Patient characteristics such as age and BMI will be compared with a two-sample T test to make sure that the two groups are equally representative.

All hemodynamic measurements such as heart rate and blood pressure will be compared with two-sample T-test. For ordinal variables such as Apgar scores and maternal nausea, a Wilcoxon-Mann Whitney test will be used. The occurrence of maternal vomiting will be compared using a Fisher's exact test.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists classification (ASA)1 and 2 patients
* non-laboring and singleton pregnancy

Exclusion Criteria:

* patients with cardiovascular comorbidities
* any kind of cardiac and peripheral vascular disease or diabetes
* history of coagulopathy
* contra-indication to spinal anesthesia
* allergic condition to vasopressors or local anesthetics
* total body weight under 50kg or above 100kg
* length under 150cm and over 180cm Body Mass Index (BM)I ≥ 32

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 11 (Actual)
Dates: Start 2022-06-09 (Actual); Primary Completion 2023-03-02 (Actual); Study Completion 2025-08-27 (Actual)

PRIMARY OUTCOMES:
dose norepinephrine used in group A | from administration of spinal anesthesia until delivery of the newborn
  dose in microgram of norepinephrine used for treatment of hypotension in both arms
dose norepinephrine used in group B | from administration of spinal anesthesia until delivery of the newborn
  dose in microgram of norepinephrine used for treatment of hypotension in both arms

SECONDARY OUTCOMES:
biochemical effect of norepinephrine on the newborn | bloodsample taken from umbilical cord at birth
  deviation of normal mean arterial pH 7.26 of the newborn

CONTACTS AND LOCATIONS:
Overall Officials: Hanne Ryckebosch, MD, Principal Investigator — University Hospital, Antwerp
Locations (1):
- Antwerp University Hospital, Edegem, Belgium